CLINICAL TRIAL: NCT02842502
Title: Clinical Feasibility of an Advanced Therapy Medicinal Product (ATMP) Preparation for Autologous Skin Regeneration in Patients Carriers of Leg Ulcers
Brief Title: Clinical Feasibility of an Advanced Therapy Medicinal Product (ATMP) Preparation for Autologous Skin Regeneration in Case of Chronic Leg Ulcers
Acronym: MecaSkin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: API/2012/33
Record Dates: First submitted 2016-07-18; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Leg Ulcer
Keywords: Skin Substitutes
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Skin graft pellet (Experimental): This group concerns patients who are recruited for skin graft procedure leading to the collection of supernumerary biopsies.
  Interventions: Procedure: Collection of supernumerary biopsies during skin graft pellet procedure

INTERVENTIONS:
Procedure: Collection of supernumerary biopsies during skin graft pellet procedure

SUMMARY:
This study deals with the feasibility of an ATMP (Advanced Therapy Medicinal Product) production for the treatment of chronic wounds ulcer. Recruitment concerns patients (n=7) with leg ulcers and receiving a skin pellet graft. During surgical procedure, supernumerary biopsies are planned to be done in order to be transferred to laboratory. Then, the possibility of cell extraction (keratinocytes and fibroblasts), expansion, banking and use for skin substitute production in clinical condition is evaluated (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic leg ulcers evolving for more than 6 months
* Patient to receive skin pellet transplant
* Chronic wound area between 10 and 30 cm²

Exclusion Criteria:

* Patient without health insurance,
* Pregnant womens,
* Smoking patient,
* Chronic wound area >30 cm²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Number of skin substitute reconstructed with cells isolated from patient biopsies | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Humbert, MD PhD, Principal Investigator — University Hospital of Besançon
Locations (1):
- CHRU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Yes